CLINICAL TRIAL: NCT01326611
Title: Efficacy of Clarithromycin Treatment in Prevention of Chronic Lung Disease in Premature Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: rö05053781128
Record Dates: First submitted 2011-03-29; First posted 2011-03-31 (Estimated); Last update posted 2011-03-31 (Estimated); Status verified 2008-05

CONDITIONS: Chronic Lung Disease
Keywords: Chronic lung disease; Clarithromycin; Ureaplasma urealyticum
MeSH Terms: interventions — Clarithromycin; Glucose

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clarithromycine Group: Active Comparator (Active Comparator): Drug: Clarithromycin intravenous clarithromycin (10 mg/kg twice a day for 10 days)
  Interventions: Drug: Clarithromycin
- Placebo Group: Placebo Comparator (Placebo Comparator): Drug: D5W Dose given daily, IV same volume that Clarithromycin would be to equal 10 mg/kg for first 10 days.
  Interventions: Drug: Dextrose

INTERVENTIONS:
Drug: Clarithromycin
  Arms: Clarithromycine Group: Active Comparator
Drug: Dextrose
  Arms: Placebo Group: Placebo Comparator

SUMMARY:
The purpose of this study is to evaluate the efficacy of clarithromycin in eradication of ureaplasma urealyticum and prevention of chronic lung disease in premature infants with birthweight < 1250 g and have ureaplasma urealyticum colonization.

ELIGIBILITY:
Inclusion Criteria:

* The babies under 1250 gram
* The babies must be appropriate for gestational age

Exclusion Criteria:

* Multiple congenital anomalies or known syndromes
* Intrauterine growth retardation with birthweight less than 10 percentile for gestational age

Ages: 1 Hour to 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 273 (Actual)
Dates: Start 2008-05; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of clarithromycin in eradication of Ureaplasma urealyticum from premature nasopharynges | 12 days after treatment by clarithromycin
  Efficacy of clarithromycin in eradication of Ureaplasma and incidence of CLD were the major outcomes of the study. Nasopharyngeal swabs for Ureaplasma were taken in postnatal first 3 days and on the 12th day only in culture positive infants, transported to the laboratory and cultured for Uu immediately.

SECONDARY OUTCOMES:
To evaluate the efficacy of clarithromycin in prevention of Chronic lung disease in premature infants with birthweight <1250 g and have Ureaplasma urealyticum colonization. | From first day of inclusion of study to at postpartum 36th week of day
  Efficacy of clarithromycin in eradication of Ureaplasma urealyticum and incidence of chronic lung disease were the major outcomes of the study. Chronic lung disease of newborn was defined as a persistent oxygen requirement at 36 weeks post menstrual age or death.

CONTACTS AND LOCATIONS:
Overall Officials: Omer Erdeve, Ass Prof, Study Director — Zekai Tahir Burak Women's Health Research and Education Hospital; Evrim Alyamac Dizdar, MD, Principal Investigator — Zekai Tahir Burak Women's Health Research and Education Hospital
Locations (1):
- Zekai Tahir Burak Maternity Teaching Hospital Neonatology department, Ankara, Turkey (Türkiye)